CLINICAL TRIAL: NCT04302259
Title: An Early Feasibility Study to Evaluate ISI-C in SCI Patients
Brief Title: Intelligent Spine Interface, Clinical (ISI-C)
Acronym: ISI-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Brown University (Other); Intel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 001020
Record Dates: First submitted 2020-02-19; First posted 2020-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SCI Patient (Experimental): Complete or Incomplete Spinal Cord Injury (SCI) patients with Asia Impairment Score (AIS) of A or B between the levels of C7/T1 and T10
  Interventions: Device: Intelligent Spine Interface

INTERVENTIONS:
Device: Intelligent Spine Interface — ISI-C is a bi-directional, two anatomical location Epidural Electrical Stimulation (EES) system to bridge the lesion core in patients with chronic complete and incomplete spinal cord injury (SCI). This "Intelligent Spine Interface", or ISI will interpret recorded neural information from above a spinal cord lesion and transfer that information, via deep neural network-based interpreters (i.e. models), to stimulation sites (electrodes) below the lesion with the aim of restoring volitional control of the lower limb.
  Other Names: spinal neuromodulation therapy, spinal cord stimulation device, epidural electrical stimulation system

SUMMARY:
This research study is being done to test a new device developed for spinal cord injury (SCI) patients. The purpose of this study is to collect data on how the nervous system signals travel within the spinal cord of SCI patients. Once the investigators understand that, they hope to develop a device that may help rehabilitation of SCI patients so that they can regain function in their lower limbs.

This study involves some imaging studies (e.g. X-rays etc.), surgical implantation of a portion of the electrical stimulation device, various assessments of body function (e.g. balance, movement, gait), and physical rehabilitation procedures. What is new and experimental is the stimulation/sensing device (Intelligent Spine Interface - Commercial, ISI-C) that will be implanted.

DETAILED DESCRIPTION:
Intel Corporation, Nuvectra 18. US FDA Regulated: Yes 19. US FDA Regulated Drug: No 20. US FDA Regulated Device: Yes 21. US FDA Investigational New Device (IND)/Investigational Device Exemption (IDE): Yes 22. Human Subjects Protection Review: Pending Review 23. Data Monitoring Committee: Yes 24. FDA Regulated Intervention: Yes

25. Brief Summary:

This research study is being done to test a new device developed for spinal cord injury (SCI) patients. The purpose of this study is to collect data on how the nervous system signals travel within the spinal cord of SCI patients. Once the investigators understand that, they hope to develop a device that may help rehabilitation of SCI patients so that they can regain function in their lower limbs.

This study involves some imaging studies (e.g. X-rays etc.), surgical implantation of a portion of the electrical stimulation device, various assessments of body function (e.g. balance, movement, gait), and physical rehabilitation procedures. What is new and experimental is the stimulation/sensing device (Intelligent Spine Interface) that will be implanted.

26. Detailed Description:

The investigators propose to build an Intelligent Spine Interface (ISI) that will interpret neural information from above a spinal cord injury and transfer that information, via a state-of-the-art artificial neural network-based computer interpreter, to sites below the site of injury and restore control of the lower limbs.

At present, activity-based therapies (physical rehabilitation) are only medical practices that can be used to enhance recovery after spinal cord injury. However, most affected patients, who fail to produce active movements voluntarily, experience minimal benefits from such therapies.

This study is being done to develop a new treatment modality for Spinal Cord Injury (SCI) patients. The purpose of this study is to collect data on how the nervous system signals travel within the spinal cord of SCI patients.

The device being used in this study is termed Intelligent Spine Interface. This device consists of: (1) surgically implanted electrode arrays placed above and below site of spinal cord injury. These arrays are connected to other device components outside the body (like "Ripple System") using specialized wires. (2) "Ripple System" collects readings from implanted electrode arrays. Together, these components are used to stimulate the spinal cord and sense any resulting nervous system signals. (3) Personal computer uses specialized software to interpret the nervous system activity.

The use of the ISI-C device in this study is considered investigational. This means the device has not yet been approved by the FDA.

The entire study should take about 7-8 months to complete.

Study Phases and Procedures:

* Screening Phase: Subject identification, consent process, eligibility review, preliminary assessments (imaging studies such as x-rays, blood work, physical/neurological exam, medical history, medication review, pregnancy test, electrocardiogram to assess heart health)
* Pre-rehabilitation Phase: baseline review of SCI related standardized outcome measures to understand if the device/treatment is producing the desired effect on the participant physical function (e.g. gait, balance, ability to walk, muscle tone/spasm, bowel function).
* Surgery: Pre-surgery testing, anesthesia administration, lead placement above and below the site of injury, wound closure and observation
* Inpatient Rehabilitation Phase: daily physical rehabilitation sessions in specialized gaits lab, neurostimulation protocol (small electrical pulses will be delivered to the implanted electrode array and any spinal cord activity will be recorded), follow-up SCI-related outcome measures review
* Surgery: same as above - surgically implanted leads will be removed
* Follow up phase: Follow-up physical and neurological exams to assess if there is a change in function since baseline

ELIGIBILITY:
Inclusion Criteria:

* • Adults (men or women) between the ages of 18 and 65 years old

  * Complete or Incomplete SCI with AIS grade of A or B between the levels of C7/T1 and T10 (level and degree of injury based on the international standards for neurological classification of SCI (ISNCSCI))
  * Focal area of SCI due to trauma
  * SCI date of injury > 1 year prior to enrollment
  * Completed prior SCI rehabilitation program
  * Ability to use both upper extremities to ambulate with a wheelchair or crutches
  * Distance between the conus medullaris and site of injury must be > 4 cm
  * The ability to participate in intensive physical therapy and research > 4 hours per day for 2 weeks
  * Must provide informed consent prior to study participation

Exclusion Criteria:

* • Presence of co-existing lower extremity neuropathy or disorders of the cauda equina

  * Presence of non-traumatic spinal cord pathology
  * Significant cognitive impairment or decreased level of consciousness
  * Presence of an intrathecal baclofen or morphine pump
  * Presence of a cardiac defibrillator or pacemaker
  * Presence of a deep brain stimulator device
  * Patient who has any contraindication to having a MRI performed
  * Severe or disabling joint contractures in the lower extremities
  * Presence of hematologic disorder or medication related coagulopathy that would preclude surgery
  * Lower extremity congenital or acquired deformities
  * Women who are pregnant or who are unwilling to use contraception during the study period
  * Body mass index > 30
  * Cardiopulmonary comorbidities that preclude participation in intensive physical therapy
  * Known or suspected patient non-compliance during the study period and at follow up
  * Patient life expectancy < 12 months
  * Presence of patient comorbidities or spinal anatomy that would preclude participation in the study per investigators' recommendation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety issues | 8 months
  Evaluate safety issues associated with the implantation and use of ISI technology i.e. frequency of device related adverse events

SECONDARY OUTCOMES:
Neurological Outcome Measures | 8 months
  Assess neurological outcomes before, during, and after ISI implantation in SCI patients via ISNCSCI evaluation
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via 6 Minute Walk Test
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via 10 minute timed walk test
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via Time Up and Go test
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via Spinal cord Injury Functional Ambulation Inventory
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via Spinal Cord Injury Quality of Life (SCI-QOL): Ambulation Short Form
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via SCI Functional Ambulatory Inventory (FAI)
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via Berg Balance Scale
Functional Outcome Measures | 8 months
  Assess functional outcomes before, during, and after ISI implantation in SCI patients via Mini-Best test

CONTACTS AND LOCATIONS:
Overall Officials: David Borton, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No